CLINICAL TRIAL: NCT03182114
Title: Hemodynamic Effects of Supine Position Versus Left Lateral Tilted Position During Cesarean Delivery: a Randomized Controlled Trial.
Brief Title: Supine Versus Left Lateral Tilted Position During Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-52-2017
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Supine Position; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine position (Placebo Comparator): the patient will receive spinal anesthesia by Bupivacaine; then she will be placed in supine position
  Interventions: Other: supine position; Drug: Bupivacaine
- Left lateral tilted position (Experimental): the patient will receive spinal anesthesia by Bupivacaine; then she will be placed in left lateral tilted position
  Interventions: Other: left lateral tilted position; Drug: Bupivacaine

INTERVENTIONS:
Other: supine position — the patient will be placed in regular supine position after spinal anesthesia
  Arms: supine position
Other: left lateral tilted position — the patient will be placed in left lateral tilted position after spinal anesthesia
  Arms: Left lateral tilted position
Drug: Bupivacaine — The patient will receive 10 mg Bupivacaine for spinal anesthesia
  Other Names: Marcaine

SUMMARY:
In this study, we will investigate the effect of left lateral tiling performed after spinal block on maternal hemodynamics compared to ordinary supine position

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Aortocaval compression is one of the theoretical mechanisms precipitating for post-spinal hypotension (PSH) for CD. Positioning of the patients in the left lateral tilted position after preforming spinal block was frequently considered a standard protocol for minimizing aortocaval compression and improve maternal hemodynamics during CD; however, the latest Cochrane database review reported that there is no adequate evidence to support any positioning protocol for prevention of PSH. Moreover, a recent study was conducted in full term pregnant women reporting no improvement in cardiac output with left lateral tilting. In this study, the effect of left lateral tiling performed after spinal block on maternal hemodynamics will be compared to ordinary supine position.

ELIGIBILITY:
Inclusion Criteria:

* full term
* singleton pregnant women
* scheduled for elective cesarean delivery

Exclusion Criteria:

* Cardiac morbidities
* hypertensive disorders of pregnancy
* peripartum bleeding
* baseline systolic blood pressure (SBP) < 100 mmHg
* body mass index > 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 80% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group

SECONDARY OUTCOMES:
severe postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 60% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group
Post-delivery hypotension | 10 minutes after delivery
  number of patients who develop hypotension (defined as decreased SBP less than 80% of the baseline reading after delivery of the fetus and starting oxytocin infusion
systolic blood pressure | 60 minutes after spinal block
  systolic blood pressure measured in mmHg
diastolic blood pressure | 60 minutes after spinal block
  diastolic blood pressure measured in mmHg
heart rate | 60 minutes after spinal block
  heart rate measured in beats per minute
incidence of nausea and vomiting | 60 minutes after spinal block
  number of patients who develop nausea and vomiting divided by the total number of patients in the group
ephedrine consumption | 60 minutes after spinal block
  total amount of ephedrine consumed during the operation (measured in milligrams)
Atropine consumption | 60 minutes after spinal block
  total amount of atropine consumed during the operation (measured in milligrams
APGAR score | 1 minute after delivery
  APGAR score for detection of the well being of the fetus
APGAR score | 10 minute after delivery
  APGAR score for detection of the well being of the fetus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Chair — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No